CLINICAL TRIAL: NCT02462512
Title: Validation of Diagnostic Performance of Ultrasound Elastography for Detection of Thyroid Cancer
Brief Title: Diagnostic Performance of Ultrasound Elastography for Detection of Thyroid Cancer
Acronym: Elastography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dong Jun Lim (Other)
Responsible Party: Sponsor-Investigator, Dong Jun Lim, SeoulStMary, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: SeoulStMary
Record Dates: First submitted 2015-04-20; First posted 2015-06-04 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Elastography; Thyroid Nodule
Keywords: Elastography; Thyroid nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FNAB of Thyroid nodule: The Patients with thyroid nodule who are scheduled for FNAB

SUMMARY:
For patients with thyroid gland nodule, fine-needle aspiration biopsy has been proved to be an efficient tool for thyroid cancer diagnosis. However, it is somewhat an invasive procedure and is subject to sampling and analysis uncertainties. Thus, improved, more reliable criteria for determining which nodule should be be aspirated are needed. Ultrasound elastography has been shown to be useful in the differential diagnosis of breast and prostate cancers. Ultrasound elastography also may discriminate malignant from benign nodule.

DETAILED DESCRIPTION:
To prospectively evaluate the elastographic appearance of thyroid cancer and explore the potential sensitivity and specificity of elastography for differentiating benign and malignant tumors, with histopathologic analysis as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

- The patients with thyroid nodule who are supposed to take fine needle aspiration biopsy

Exclusion Criteria:

- The patients who do not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with thyroid nodule who visit tertiary hospital for fine needle aspiration biopsy
Sampling Method: Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of elastography using in-vivo compression for detection of thyroid cancer | 1 year
  Measuring ECI(Elasticity contrast index) of thyroid nodule by ultrasound elastography

SECONDARY OUTCOMES:
Determination of the parameters which could have influence on the diagnostic performance of ultrasound elastography using in-vivo compression | One year
  Analysis of clinical characteristics of thyroid nodules and patients which are related to the diagnostic performance of ultrasound elastography

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jun Lim, Dr., Principal Investigator — Associate Professor, Head, Division of Endocrinology and Metabolism, Department of Internal Medicine, College of Medicine, The Catholic University of Korea; Min Hee Kim, Dr., Study Director — Clinical Assistant Professor, Division of Endocrinology and Metabolism, Department of Internal Medicine, College of Medicine, The Catholic University of Korea
Locations (1):
- Seoul St Mary's Hospital, Seocho-gu, Seoul, South Korea

REFERENCES:
- [Background] Dighe M, Bae U, Richardson ML, Dubinsky TJ, Minoshima S, Kim Y. Differential diagnosis of thyroid nodules with US elastography using carotid artery pulsation. Radiology. 2008 Aug;248(2):662-9. doi: 10.1148/radiol.2482071758. Epub 2008 Jun 6. PMID 18539888
- [Result] Luo S, Lim DJ, Kim Y. Objective ultrasound elastography scoring of thyroid nodules using spatiotemporal strain information. Med Phys. 2012 Mar;39(3):1182-9. doi: 10.1118/1.3679857. PMID 22380349
- [Result] Lim DJ, Luo S, Kim MH, Ko SH, Kim Y. Interobserver agreement and intraobserver reproducibility in thyroid ultrasound elastography. AJR Am J Roentgenol. 2012 Apr;198(4):896-901. doi: 10.2214/AJR.11.7009. PMID 22451558